CLINICAL TRIAL: NCT00072722
Title: Phase II Randomized Open-Label, Two-Arm Study of Safety and Efficacy of CC-4047 in Subjects With Metastatic Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Safety and Efficacy of CC-4047 in Subjects With Metastatic Hormone Refractory Prostate Cancer (HRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-PC-002
Record Dates: First submitted 2003-11-07; First posted 2003-11-13 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Metastatic Hormone Refractory Prostate Cancer; CC4047; CC-4047; Prostate Carcinoma; Celgene
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pomalidomide

INTERVENTIONS:
Drug: CC-4047

SUMMARY:
Phase II randomized open-label, two-arm study of safety and efficacy of CC-4047 in subjects with metastatic hormone refractory prostate cancer (HRPC)

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Adult male subjects, age 18 or older at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Histologically confirmed adenocarcinoma of the prostate with radiographic evidence of metastases and PSA progression following hormonal therapy for metastatic disease. Subjects must have evidence of progression of disease as demonstrated by 2 consecutive rises in PSA (an absolute change of at least 1ng/ml) separated by at least 28 days.
* Antiandrogen therapy must have been stopped at least 4 weeks (for flutamide) or 6 weeks (for bicalutamide or nilutamide) prior to entering study with evidence of a rising PSA (from baseline) measured x 2 at least 2 weeks apart Testicular androgen suppression must be maintained with either LHRH therapy of bilateral orchiectomy.
* Must use barrier contraception (latex condom) when engaging in reproductive activity with women of child-bearing potential throughout the course of study treatment and for 4 weeks following the discontinuation of study treatment.
* May have had only one prior regimen of chemotherapy for prostate cancer. The chemotherapy must have been stopped at least 4 weeks prior to study entry.
* Disease-free of other malignancies for greater than 5 years with the exception of curatively treated basal cell, squamous cell carcinoma of the skin of Ta transitional cell carcinoma of the bladder.
* ECOG performance status of 0 or 1.
* Serum creatinine greater than or equal to 2.0 mg%
* Adequate hematologic functions: Granulocytes greater than or equal to 1800 mm3 and platelets greater than or equal to 100,000 mm3.
* Adequate hepatocellular function: AST<2 x normal and bilirubin<1.5mg/dl
* No active unresolved infection

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Any prior use of CC-4047 of Thalidomide
* Tumors containing small cell or sarcomatoid elements
* Symptomatic bone metastases.
* Concurrent use of any other anti-cancer agents.
* Known brain disease that is symptomatic, is currently being treated with corticosteroids, or has not been previously irradiated.
* Non-PSA producing tumors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-09; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Health Science Center, Denver, Colorado
  - Baylor College of Medicine, Houston, Texas